CLINICAL TRIAL: NCT06013332
Title: A Controlled, Randomized, Double-Blinded, Intra-Subject, Multicenter, Prospective, Clinical Study to Investigate the Non-Inferiority Between the Polymeric Microspheres and Sculptra® in the Treatment of Moderate to Severe Nasolabial Folds
Brief Title: Polymeric Microspheres vs Sculptra® in the Treatment of Moderate to Severe Nasolabial Folds
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Hospital (Other)
Collaborators: Taipei Medical University (Other); Panion & BF Biotech Inc. (Industry)
Responsible Party: Principal Investigator, Hsiou-Hsin Tsai, Visiting Staff, Taipei Medical University Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PBF-PLLA-001
Record Dates: First submitted 2023-08-13; First posted 2023-08-28 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Nasolabial Fold Wrinkles

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): right face will be injected with PBF PLLA microsphere, and left face with Sculptra®
  Interventions: Device: PBF PLLA microsphere (injectable poly-L-lactic acid); Device: Sculptra®
- Group 2 (Experimental): right face will be injected with Sculptra® and left face with PBF PLLA microsphere
  Interventions: Device: PBF PLLA microsphere (injectable poly-L-lactic acid); Device: Sculptra®

INTERVENTIONS:
Device: PBF PLLA microsphere (injectable poly-L-lactic acid) — Poly-L-lactic acid (PLLA) is a collagen stimulator, helps restore the deep, underlying structure of the skin to diminish facial wrinkles. PLLA microparticles are absorbable for human body, and it works with human body within the deep dermis to help revitalize collagen production and help restore human skin's inner structure and volume. PLLA can rebuilt collagen strands begin gradually helping to restore facial volume and the look of fullness to wrinkles and folds.
Device: Sculptra® — Sculptra®

SUMMARY:
This is a single-dose, randomized, double-blind, active-controlled, split-face, multiple centers, non-inferiority study. Approximately 50 nasolabial fold subjects will be enrolled. Each enrolled subject will be randomized equally into one of the following groups:

1. Group 1: right face will be injected with PBF PLLA microsphere, and left face with Sculptra®
2. Group 2: right face will be injected with Sculptra® and left face with PBF PLLA microsphere Subjects will be administrated on Visit 1 by applying PBF PLLA microsphere on one side of face and Sculptra® on the other.

ELIGIBILITY:
Inclusion Criteria:

1. Participant whose age is ≥ 18 and ≤ 65 years old.
2. Participant who is able to read, understand, sign, and date a written informed consent form (ICF) before study participation at screening.
3. Participant is able to understand and comply with protocol requirements and instructions and likely to complete the study as planned.
4. Participant who has moderate to severe nasolabial folds on two sides of face, WAS Score ≥ 3. WAS Score is determined by investigator.
5. Participant whose difference in WAS score of nasolabial folds on two sides of face ≤ 1. WAS Score is determined by investigator.
6. Participant's skin condition is considered by Investigator suitable for the treatment of Poly-L-lactic Acid (PLLA).

Exclusion Criteria:

-

1. Participant who has previous tissue augmenting therapy, contouring or revitalization treatment in or near the treatment area prior to the Baseline visit.

1. Treatment with collagen or hyaluronic acid (HA) in the last 12 months.
2. Had facelift treatment (high intensity focused ultrasound, radio frequency, or thread) within 12 months.
3. Had face laser treatment within 6 months.
4. Had been treated with Calcium Hydroxyapatite (CaHA), PLLA or permanent (non-biodegradable).

2. Participant who has severe allergies with a history of severe reactions (anaphylaxis) or multiple severe allergies or has known/previous allergy or hypersensitivity to any of the PLLA, other constituents of PBF PLLA microsphere or Sculptra®, or drugs containing lidocaine such as Lidiprine Cream and its constituents. 3. Participant who has obvious defects, trauma, or scars near the treatment area.

4. Participant who has been diagnosed head cancer in the last 3 years. 5. Participant who has trauma, open wound, active skin disease or inflammation at the injection site.

6. Participant who has serious systematic disease that judged by Investigator which is not suitable for the treatment.

7. Participant who has connective tissue disease, bleeding disorders, active hepatitis, immune deficiency disease, disease such as cancer, stroke and/or myocardial infarction and on any immunosuppressive therapy.

8. Participant who previously had or have risks factors for hypertrophic scarring or keloid formation near the treatment area.

9. Participant who has used immune system suppression drugs, steroids, anti-inflammatory drugs, anticoagulant drugs, or aspirin within 7 days before treatment.

10. Female participant who is pregnant or lactating.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Delta of the WAS score between the Baseline and 26 weeks after treatment assessed by the Independent Evaluators of PLLA(PBF) versus Sculptra® | 26 weeks
  Wrinkle Assessment Scale (WAS): 0 No wrinkles; 1 Just perceptible wrinkle; 2 Shallow wrinkles; 3 Moderately deep wrinkle; 4 deep wrinkle, well-defined edges; 5 Very deep wrinkle, redundant fold

SECONDARY OUTCOMES:
Overall operation time during subcutaneous injection of PLLA(PBF) versus Sculptra® | First week from the Start of administration to the end of administration
  To compare the operational smoothness for physicians between the two medical devices
Delta of the WAS score assessed by the Investigator between each follow-up visit (13th, 26th, 39th and 52nd week post-administration) and the Baseline of PLLA(PBF) versus Sculptra® | 13th, 26th, 39th and 52nd week post-administration
  Wrinkle Assessment Scale (WAS): 0 No wrinkles; 1 Just perceptible wrinkle; 2 Shallow wrinkles; 3 Moderately deep wrinkle; 4 deep wrinkle, well-defined edges; 5 Very deep wrinkle, redundant fold
Delta of the WSRS score between the Baseline and 26 weeks after treatment assessed by the Independent Evaluators of PLLA(PBF) versus Sculptra® | 26 weeks
  Grade 1: No visible nasolabial fold; continuous skin line Grade 2: Shallow but visible nasolabial fold with a slight indentation; minor facial feature; the implant is expected to produce a slight improvement in appearance Grade 3: Moderately deep nasolabial folds; clear facial feature visible at normal appearance but not when stretched; excellent correction is expected with injectable implant Grade 4: Very long and deep nasolabial folds; prominent facial feature; 2mm visible fold when stretched; significant improvement is expected with injectable implant Grade 5: Extremely deep and long nasolabial folds, detrimental to facial appearance; 2-4mm visible V-shaped fold when stretched; unlikely to have satisfactory correction with injectable implant alone
Delta of the WSRS score assessed by the Investigator between each follow-up visit (13th, 26th, 39th and 52nd week post-administration) and the Baseline of PLLA(PBF) versus Sculptra® | 13th, 26th, 39th and 52nd week post-administration
  Grade 1: No visible nasolabial fold; continuous skin line Grade 2: Shallow but visible nasolabial fold with a slight indentation; minor facial feature; the implant is expected to produce a slight improvement in appearance Grade 3: Moderately deep nasolabial folds; clear facial feature visible at normal appearance but not when stretched; excellent correction is expected with injectable implant Grade 4: Very long and deep nasolabial folds; prominent facial feature; 2mm visible fold when stretched; significant improvement is expected with injectable implant Grade 5: Extremely deep and long nasolabial folds, detrimental to facial appearance; 2-4mm visible V-shaped fold when stretched; unlikely to have satisfactory correction with injectable implant alone
Percentage of responders based on the intra-individual improvement of at least one grade in the WAS score compared to baseline assessed by the Investigator of PLLA(PBF) versus Sculptra® | 13th, 26th, 39th and 52nd week post-administration
  Wrinkle Assessment Scale (WAS): 0 No wrinkles; 1 Just perceptible wrinkle; 2 Shallow wrinkles; 3 Moderately deep wrinkle; 4 deep wrinkle, well-defined edges; 5 Very deep wrinkle, redundant fold
Percentage of responders based on the intra-individual improvement of at least one grade in the WSRS score compared to baseline assessed by the Investigator of PLLA(PBF) versus Sculptra® | 13th, 26th, 39th and 52nd week post-administration
  Grade 1: No visible nasolabial fold; continuous skin line Grade 2: Shallow but visible nasolabial fold with a slight indentation; minor facial feature; the implant is expected to produce a slight improvement in appearance Grade 3: Moderately deep nasolabial folds; clear facial feature visible at normal appearance but not when stretched; excellent correction is expected with injectable implant Grade 4: Very long and deep nasolabial folds; prominent facial feature; 2mm visible fold when stretched; significant improvement is expected with injectable implant Grade 5: Extremely deep and long nasolabial folds, detrimental to facial appearance; 2-4mm visible V-shaped fold when stretched; unlikely to have satisfactory correction with injectable implant alone
Number of subjects scored either 'Much Improved' or 'Improved' on GAIS evaluated by the Investigator for PLLA(PBF) versus Sculptra® | 13th, 26th, 39th and 52nd week post-administration
Subject's satisfaction score (Subjective 5-point scale with 1 being 'very satisfied' and 5 being 'very dissatisfied') of PLLA(PBF) versus Sculptra® | 13th, 26th, 39th and 52nd week post-administration

OTHER OUTCOMES:
Post injection treatment responses (From common treatment responses diary card) for safety evaluation of PBF PLLA microsphere versus Sculptra® | During 2 weeks post-administration
Assessment of injection site pain of PBF PLLA microsphere versus Sculptra® by using Visual Analogue Scale (VAS) score | immediately after injection and at 5-, 15- and 30- minute post-administration
Compare the treatment related adverse event | During 52 weeks post-administration

CONTACTS AND LOCATIONS:
Overall Officials: Hsiou-Hsin Tsai, M.D. PhD., Principal Investigator — Taipei Medical University Hospital
Locations (2):
- Taiwan (2):
  - Taipei Medical University Hospital, Taipei
  - Taipei Municipal Wanfang Hospital, Taipei